CLINICAL TRIAL: NCT03742180
Title: A Prospective Randomized Trial of Sublingual Ketorolac Compared to Intranasal Dexmedetomidine for Postoperative Analgesia in Pediatric Patients Undergoing Bilateral Myringotomy
Brief Title: Sublingual Ketorolac Compared to Intranasal Dexmedetomidine for Postoperative Analgesia in Pediatric Patients Undergoing Bilateral Myringotomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unavailable drug in Egypt.
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R/18.06.212
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Elective Bilateral Myringotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal dexmedetomidine (Experimental): this group is planned for intranasal dexmedetomidine
  Interventions: Drug: intranasal dexmedetomidine
- sublingual ketorolac (Active Comparator): this group is planned for sublingual ketorolac
  Interventions: Drug: sublingual ketorolac

INTERVENTIONS:
Drug: intranasal dexmedetomidine — The patient will receive intranasal dexmedetomidine in a dose of 1ug.kg-1 in a volume of 1 ml was dripped into both nostrils using a 1-mL syringe, with the patients in the recumbent position plus 1ml sublingual 0.9% saline
  Arms: intranasal dexmedetomidine
Drug: sublingual ketorolac — The patient will receive sublingual ketorolac in a dose of 0.5 mg.kg-1 in a volume of 1 ml and 1 ml intranasal saline 0.9%
  Arms: sublingual ketorolac

SUMMARY:
The investigators aim to compare intranasal dexmedetomidine in a dose of 1ug.kg-1 with sublingual ketorolac in a dose of 1mg.kg-1 on postoperative behaviour in those children undergoing BMT during their PACU stay

DETAILED DESCRIPTION:
Data were analyzed through SPSS (Statistical Package for Social Sciences), Program version 22. Distribution of data was first tested by Shapiro test. Data were presented as the mean and standard deviation (SD), median and range or numbers and percentages. For normally distributed data, an unpaired t-test was used to compare between mean values of both groups. For pain and sedation scores, Mann Whitney U test was used. Fisher's exact test was used for comparison of categorical data. The P value ≤ 0.05 was considered as the level of statistical significance.

A prior G power analysis was done. Using the results obtained from previous studies (14- 18) and assuming an alpha error of 0.05 and beta error 0f 0.2 (power of the study 80 %), a sample size of 60 patients per group was calculated. A drop out 10% of cases is expected, so; 33 cases per group will be required

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I- II.

Exclusion Criteria:

* History of ketamine
* History of NSAID
* History of allergies
* Any bleeding disorders
* History of GIT bleeding
* Those who will undergo other procedures in addition to bilateral myringotomy

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | time from administering the study solution till the time for the first rescue analgesic] during first 24 hours
  The duration of analgesia,define as the time to the first demand for rescue analgesic

SECONDARY OUTCOMES:
Postoperative pain score | For 24 hours after surgery
  Postoperative pain will be assessed by the CHEOP scale (Children's Hospital of Eastern Ontario Pain Scale) .
Heart rate | for 2 hours after the start of surgery
systolic blood pressure | for 2 hours after the start of surgery
Number of patients received rescue analgesics | For 24 hours after surgery
  Total number of children who required postoperative pain medication during the 24-h period will be registered
Degree of sedation | For 24 hours after surgery
  The degree of sedation will be assessed by using Ramsay scale
Nausea and vomiting | For 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided